CLINICAL TRIAL: NCT06967142
Title: Fluid Responsiveness Through the Corrected Carotid Flow Time, Before and After Sternotomy
Status: Completed | Type: Observational
Sponsor: Ankara City Hospital Bilkent (Other)
Responsible Party: Principal Investigator, Seda Kurtbeyoğlu, Principal Investigator, doctor, Ankara City Hospital Bilkent
Other Study IDs: Corrected Carotid Flow Time
Record Dates: First submitted 2025-03-02; First posted 2025-05-13 (Actual); Last update posted 2025-05-18 (Actual); Status verified 2025-05

CONDITIONS: Coronary Artery Disease
Keywords: corrected carotid flow time; fluid responsiveness
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Study group: The study was conducted at the Cardiovascular Surgery Operating Room of the Ministry of Health Ankara Bilkent City Hospital. Fifty patients, aged 18-80 years, classified as ASA II-III, who were scheduled for elective coronary artery bypass graft surgery under general anesthesia, were included in the study. Three patients were excluded due to missing data, and two patients were excluded due to hemodynamic instability, leaving 45 patients in total.
  Hemodynamic parameters, including heart rate (HR) (beats/min), central venous pressure (CVP, mmHg), systolic arterial blood pressure (SAB, mmHg), diastolic arterial blood pressure (DAB, mmHg), mean arterial pressure (MAP, mmHg), stroke volume index (SVI), cardiac index (CI), PPV, SVV, and carotid artery FTc, were assessed and recorded six times:
  1.before sternotomy and 2.after LRM, 3.after sternotomy and 4.after LRM, 5.before and 6.after fluid loading
  Interventions: Device: Correcte Carotid flow measurement by USG Doppler

INTERVENTIONS:
Device: Correcte Carotid flow measurement by USG Doppler — Aim of this study is to investigate the usability of changes in corrected carotid flow time induced by lung recruitment maneuvers during protective lung ventilation (6 ml/kg tidal volume) in patients undergoing elective Coronary Artery Bypass Graft Surgery (CABG) to evaluate fluid responsiveness. The secondary objective is to determine the correlation between measurements taken before and after sternotomy. This study aims to reduce invasive procedures used for assessing fluid responsiveness and develop an alternative method to the use of hard-to-access devices for measurements.

SUMMARY:
Perioperative fluid management is used to maintain the perfusion of vital organs, prevent hypovolemia, inadequate tissue perfusion, and tissue edema, and cardiovascular complications caused by the infusion of large amounts of blood and blood products. Optimal fluid management improves postoperative outcomes. However, excessive or inadequate fluid infusion increases morbidity. Traditional fluid therapy strategies are divided into three groups: liberal fluid therapy, restrictive fluid therapy, and goal-directed therapy (GDT).

Fluid responsiveness refers to a patient's hemodynamic response to intravenous fluid loading and is defined as an increase of 10% or more in stroke volume (SV) or cardiac output (CO). Various parameters are used to assess fluid responsiveness. Static parameters have limited accuracy in predicting fluid responsiveness. Dynamic parameters such as stroke volume variation (SVV), pulse pressure variation (PPV), passive leg raising test (PLR), and end-expiratory occlusion test (EEOT) have been found to be more reliable in assessing fluid responsiveness.

The pulse contour analysis method (PCA) continuously measures cardiac output by analyzing the arterial pressure waveform. The ProAQT/PulsioFlex system measures cardiac output by analyzing the arterial waveform without requiring calibration.

Lung recruitment maneuvers (LRM) are techniques used in mechanically ventilated patients to prevent atelectasis and improve oxygenation. They have also been shown to assist in assessing fluid responsiveness. LRM methods include sustained inflation (SI), increased PEEP pressure, increased tidal volume, and targeted recruitment. The temporary increase in intrathoracic pressure during LRM can affect stroke volume variation and be used to assess fluid responsiveness.

Corrected carotid flow time (FTc) is a non-invasive parameter calculated by normalizing the systolic ejection time in the carotid artery to heart rate. FTc can be measured using Doppler ultrasound. It is thought that changes in FTc measured during passive leg raising (PLR) or lung recruitment maneuvers (LRM) may help identify fluid-responsive patients, and new studies are being conducted on this topic.

Recent studies suggest that changes in FTc during lung recruitment maneuvers may be a reliable method for assessing fluid responsiveness.

The optimal method for assessing fluid responsiveness during lung-protective ventilation remains unknown. In patients who have undergone sternotomy with an open chest wall, an ideal method for evaluating fluid responsiveness has not yet been determined.

The primary objective of this study is to investigate the usability of changes in corrected carotid flow time induced by lung recruitment maneuvers during protective lung ventilation (6 ml/kg tidal volume) in patients undergoing elective Coronary Artery Bypass Graft (CABG) surgery to evaluate fluid responsiveness. The secondary objective is to determine the correlation between measurements taken before and after sternotomy. This study aims to reduce invasive procedures used for assessing fluid responsiveness and minimize the need for difficult-to-access devices for measurements.

The study was conducted in the Cardiovascular Surgery Operating Room at the Ministry of Health Ankara Bilkent City Hospital. Fifty patients, aged 18-80 years, classified as ASA II-III, who were scheduled for elective coronary artery bypass graft surgery under general anesthesia, were included in the study. Three patients were excluded due to missing data, and two patients were excluded due to hemodynamic instability, leaving 45 patients in total. The study was designed as a single-center, prospective, observational study and was conducted between July 1, 2024, and November 1, 2024.

All patients included in the study were monitored in the same standard way. Heart rate, intra-arterial monitoring, and PulsioFlex monitoring were performed. All patients were given the same induction and anesthesia maintenance. Fluid responsiveness was evaluated by measurements taken at specific intraoperative times. Hemodynamic parameters, including heart rate (HR) (beats/min), central venous pressure (CVP, mmHg), systolic arterial blood pressure (SAB, mmHg), diastolic arterial blood pressure (DAB, mmHg), mean arterial pressure (MAP, mmHg), stroke volume index (SVI), cardiac index (CI), PPV, SVV, and carotid artery FTc, were assessed and recorded six times:

T1:After induction is complete and preparations are made for the surgical procedure, before incision is started T2:Before starting sternotomy, 1 minute after LRM T3:After sternotomy within 5 minutes T4:After sternotomy, LRM is applied when hemodynamic stability is achieved. Measurement is made 1 minute after LRM.

T5:Measurement is made 10 minutes after T4 when hemodynamic parameters are stable.

T6:After the T5 measurement, the patient All measurements were taken at the beginning of surgery, terminated after 12 hours from the induction .

DETAILED DESCRIPTION:
Measurements will be taken six times:

T1.Before sternotomy T2.After LRM is performed before sternotomy T3.5 minutes After sternotomy T4.LRM was performed 10 minutes after sternotomy, the recording will be taken within 2 minutes after the LRM is finished T5.Before fluid loading (15 minutes after T4 if hemodynamics are stable) T6.After fluid loading (After the T5 measurement is taken, the fluid loading is done and after the fluid is finished, within 2 minutes T6 measurement is taken) We expect these measurements to be made during the first half of the surgery; if for any reason it takes longer than 12 hours, the patient will be removed from study

ELIGIBILITY:
Inclusion Criteria:

* ASA 2-3 patients
* Aged 18-80 years
* Will undergo elective coronary bypass surgery under general anesthesia

Exclusion Criteria:

* Age <18 or >80 years
* Patients with an ASA score greater than 3
* Ejection fraction (EF) <40%
* Patients with contraindications to anesthetic drugs
* BMI >30
* Patients who do not wish to participate in the study
* Right ventricular dysfunction
* Chronic obstructive pulmonary disease (COPD)
* Bullous lung disease
* Moderate to severe pulmonary hypertension (PHT)
* Severe renal or liver disease
* Patients who develop hemodynamic instability in the perioperative period
* Pregnancy

Criteria for Study Termination:

* Patients who develop hemodynamic instability during LRM
* Patients who experience unexpected intraoperative surgical complications

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: ASA 2-3 patients aged 18-80 years who will undergo elective coronary bypass surgery under general anesthesia in the cardiovascular surgery operating room of Ankara City Hospital.
Sampling Method: Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2025-01-01 (Actual); Primary Completion 2025-02-25 (Actual); Study Completion 2025-02-28 (Actual)

PRIMARY OUTCOMES:
corrected carotid flow time | 12 hours
  The corrected carotid flow time (ccFT) was measured using Doppler ultrasound. The USG probe is placed on the carotid artery and the carotid flow wave is recorded.
  CFT is the duration from the beginning of the systolic waveform to the dicrotic notch and corrected for heart rate using Wodey's formula to obtain the ccFT in milliseconds (ms): Corrected carotid flow time (ccFT) = carotid flow time + 1.29 (heart rate-60).
  Measurements will be taken six times:
  T1.Before sternotomy T2.After LRM is performed before sternotomy T3.5 minutes After sternotomy T4.LRM was performed 10 minutes after sternotomy, the recording will be taken within 2 minutes after the LRM is finished T5.Before fluid loading (15 minutes after T4 if hemodynamics are stable) T6.After fluid loading (After the T5 measurement is taken, the fluid loading is done and after the fluid is finished, within 2 minutes T6 measurement is taken) We expect these measurements to be made during the first half of the surgery; if for any re
Systolic arterial blood pressure | 12 hours
  Intra-arterial cannulation and monitoring were established before the induction started. Systolic arterial blood pressure was measured and recorded as mmHg. Measurements will be taken six times:
  T1.Before sternotomy T2.After LRM is performed before sternotomy T3.5 minutes After sternotomy T4.LRM was performed 10 minutes after sternotomy, the recording will be taken within 2 minutes after the LRM is finished T5.Before fluid loading (15 minutes after T4 if hemodynamics are stable) T6.After fluid loading (After the T5 measurement is taken, the fluid loading is done and after the fluid is finished, within 2 minutes T6 measurement is taken) We expect these measurements to be made during the first half of the surgery; if for any reason it takes longer than 12 hours, the patient will be removed from study

SECONDARY OUTCOMES:
diastolic arterial blood pressure | 12 hours
  Intra-arterial cannulation and monitoring were established before the induction started. Diastolic arterial blood pressure was measured and recorded as mmHg. Measurements will be taken six times:
  T1.Before sternotomy T2.After LRM is performed before sternotomy T3.5 minutes After sternotomy T4.LRM was performed 10 minutes after sternotomy, the recording will be taken within 2 minutes after the LRM is finished T5.Before fluid loading (15 minutes after T4 if hemodynamics are stable) T6.After fluid loading (After the T5 measurement is taken, the fluid loading is done and after the fluid is finished, within 2 minutes T6 measurement is taken) We expect these measurements to be made during the first half of the surgery; if for any reason it takes longer than 12 hours, the patient will be removed from study
mean arterial blood pressure | 12 hours
  Intra-arterial cannulation and monitoring were established before the induction started. Mean arterial blood pressure was measured and recorded as mmHg. Measurements will be taken six times:
  T1.Before sternotomy T2.After LRM is performed before sternotomy T3.5 minutes After sternotomy T4.LRM was performed 10 minutes after sternotomy, the recording will be taken within 2 minutes after the LRM is finished T5.Before fluid loading (15 minutes after T4 if hemodynamics are stable) T6.After fluid loading (After the T5 measurement is taken, the fluid loading is done and after the fluid is finished, within 2 minutes T6 measurement is taken) We expect these measurements to be made during the first half of the surgery; if for any reason it takes longer than 12 hours, the patient will be removed from study
Anaesthesia debpt based on Bispectral İndex | 12 hours
  Anesthesia depth was assessed using BIS (bispectral index) monitoring during surgery and recorded . A numeric value is recorded in the range of 0-100.
  Measurements will be taken six times:
  T1.Before sternotomy T2.After LRM is performed before sternotomy T3.5 minutes After sternotomy T4.LRM was performed 10 minutes after sternotomy, the recording will be taken within 2 minutes after the LRM is finished T5.Before fluid loading (15 minutes after T4 if hemodynamics are stable) T6.After fluid loading (After the T5 measurement is taken, the fluid loading is done and after the fluid is finished, within 2 minutes T6 measurement is taken) We expect these measurements to be made during the first half of the surgery; if for any reason it takes longer than 12 hours, the patient will be removed from study
heart rate | 12 hours
  ECG monitoring was performed on the patient, and heart rate was recorded as a numeric value per second.
  Measurements will be taken six times:
  T1.Before sternotomy T2.After LRM is performed before sternotomy T3.5 minutes After sternotomy T4.LRM was performed 10 minutes after sternotomy, the recording will be taken within 2 minutes after the LRM is finished T5.Before fluid loading (15 minutes after T4 if hemodynamics are stable) T6.After fluid loading (After the T5 measurement is taken, the fluid loading is done and after the fluid is finished, within 2 minutes T6 measurement is taken) We expect these measurements to be made during the first half of the surgery; if for any reason it takes longer than 12 hours, the patient will be removed from study
Systemic vascular resistance | 12 hours
  Hemodynamic monitoring was performed on the patient with PulsionFlex, and the SVR (Systemic Vascular Resistance) value was observed as a numeric value dynes/sec/cm-5. (Normal SVR is between 900 and 1440 dynes/sec/cm-5)
  Measurements will be taken six times:
  T1.Before sternotomy T2.After LRM is performed before sternotomy T3.5 minutes After sternotomy T4.LRM was performed 10 minutes after sternotomy, the recording will be taken within 2 minutes after the LRM is finished T5.Before fluid loading (15 minutes after T4 if hemodynamics are stable) T6.After fluid loading (After the T5 measurement is taken, the fluid loading is done and after the fluid is finished, within 2 minutes T6 measurement is taken) We expect these measurements to be made during the first half of the surgery; if for any reason it takes longer than 12 hours, the patient will be removed from study
stroke volume index | 12 hours
  Hemodynamic monitoring was performed on the patient with PulsionFlex, and the SVI (stroke volume index) value was observed as a numeric value mL/m2. (Normal SVI is between 35-65mL/m2)
  Measurements will be taken six times:
  T1.Before sternotomy T2.After LRM is performed before sternotomy T3.5 minutes After sternotomy T4.LRM was performed 10 minutes after sternotomy, the recording will be taken within 2 minutes after the LRM is finished T5.Before fluid loading (15 minutes after T4 if hemodynamics are stable) T6.After fluid loading (After the T5 measurement is taken, the fluid loading is done and after the fluid is finished, within 2 minutes T6 measurement is taken) We expect these measurements to be made during the first half of the surgery; if for any reason it takes longer than 12 hours, the patient will be removed from study
cardiac index | 12 hours
  Hemodynamic monitoring was performed on the patient with PulsionFlex, and the CI (cardiac index) value was observed as a numeric value L/min/m2. (Normal CI is between 2.6 and 4.2 L/min/m2)
  Measurements will be taken six times:
  T1.Before sternotomy T2.After LRM is performed before sternotomy T3.5 minutes After sternotomy T4.LRM was performed 10 minutes after sternotomy, the recording will be taken within 2 minutes after the LRM is finished T5.Before fluid loading (15 minutes after T4 if hemodynamics are stable) T6.After fluid loading (After the T5 measurement is taken, the fluid loading is done and after the fluid is finished, within 2 minutes T6 measurement is taken) We expect these measurements to be made during the first half of the surgery; if for any reason it takes longer than 12 hours, the patient will be removed from study
Pulse Pressure Variation | 12 hours
  Hemodynamic monitoring was performed on the patient with PulsionFlex, and the PPV (Pulse Pressure Variation) value was observed as a numeric value mm Hg. Normal PPV is between 40 and 60 mm Hg)
  Measurements will be taken six times:
  T1.Before sternotomy T2.After LRM is performed before sternotomy T3.5 minutes After sternotomy T4.LRM was performed 10 minutes after sternotomy, the recording will be taken within 2 minutes after the LRM is finished T5.Before fluid loading (15 minutes after T4 if hemodynamics are stable) T6.After fluid loading (After the T5 measurement is taken, the fluid loading is done and after the fluid is finished, within 2 minutes T6 measurement is taken) We expect these measurements to be made during the first half of the surgery; if for any reason it takes longer than 12 hours, the patient will be removed from study
Stroke Volüme Variation | 12 hours
  Hemodynamic monitoring was performed on the patient with PulsionFlex, and the SVV (Stroke Volüme Variation) value was observed as a numeric value of percentage (%). The normal range of SVV under controlled ventilation is less than 10-13%.
  Measurements will be taken six times:
  T1.Before sternotomy T2.After LRM is performed before sternotomy T3.5 minutes After sternotomy T4.LRM was performed 10 minutes after sternotomy, the recording will be taken within 2 minutes after the LRM is finished T5.Before fluid loading (15 minutes after T4 if hemodynamics are stable) T6.After fluid loading (After the T5 measurement is taken, the fluid loading is done and after the fluid is finished, within 2 minutes T6 measurement is taken) We expect these measurements to be made during the first half of the surgery; if for any reason it takes longer than 12 hours, the patient will be removed from study
central venous pressure | 12 hours
  The central venous pressure was measured by a central venous catheter placed through internal jugular veins, using a pressure transducer and observed as a numeric value as mmHg. Normal CVP is approximately 2 to 8 mm Hg. Measurements will be taken six times:
  T1.Before sternotomy T2.After LRM is performed before sternotomy T3.5 minutes After sternotomy T4.LRM was performed 10 minutes after sternotomy, the recording will be taken within 2 minutes after the LRM is finished T5.Before fluid loading (15 minutes after T4 if hemodynamics are stable) T6.After fluid loading (After the T5 measurement is taken, the fluid loading is done and after the fluid is finished, within 2 minutes T6 measurement is taken) We expect these measurements to be made during the first half of the surgery; if for any reason it takes longer than 12 hours, the patient will be removed from study
Oxygen delivery | 12 hours
  Hemodynamic monitoring was performed on the patient with PulsionFlex, and the DO2 (Oxygen delivery) value was observed as a numeric value as ml/min/m2. Normal DO2 is approximately 600 ml/min/m2.
  Measurements will be taken six times:
  T1.Before sternotomy T2.After LRM is performed before sternotomy T3.5 minutes After sternotomy T4.LRM was performed 10 minutes after sternotomy, the recording will be taken within 2 minutes after the LRM is finished T5.Before fluid loading (15 minutes after T4 if hemodynamics are stable) T6.After fluid loading (After the T5 measurement is taken, the fluid loading is done and after the fluid is finished, within 2 minutes T6 measurement is taken) We expect these measurements to be made during the first half of the surgery; if for any reason it takes longer than 12 hours, the patient will be removed from study

CONTACTS AND LOCATIONS:
Overall Officials: Seda Kurtbeyoğlu, doctor, Study Director — Ankara City Hospital Bilkent; Rahime Güney, doctor, Principal Investigator — Ankara City Hospital Bilkent
Locations (1):
- Ankara Bilkent City Hospital, Çankaya, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Kimura A, Suehiro K, Juri T, Tanaka K, Mori T. Changes in corrected carotid flow time induced by recruitment maneuver predict fluid responsiveness in patients undergoing general anesthesia. J Clin Monit Comput. 2022 Aug;36(4):1069-1077. doi: 10.1007/s10877-021-00736-7. Epub 2021 Jun 30. PMID 34191254
- [Result] Lagier D, Fischer F, Fornier W, Fellahi JL, Colson P, Cholley B, Jaber S, Baumstarck K, Guidon C; PROVECS investigators and the ARCOTHOVA group. A perioperative surgeon-controlled open-lung approach versus conventional protective ventilation with low positive end-expiratory pressure in cardiac surgery with cardiopulmonary bypass (PROVECS): study protocol for a randomized controlled trial. Trials. 2018 Nov 13;19(1):624. doi: 10.1186/s13063-018-2967-y. PMID 30424770
- [Result] Watanabe R, Suehiro K, Mukai A, Tanaka K, Yamada T, Mori T, Nishikawa K. Changes in stroke volume induced by lung recruitment maneuver can predict fluid responsiveness during intraoperative lung-protective ventilation in prone position. BMC Anesthesiol. 2021 Dec 2;21(1):303. doi: 10.1186/s12871-021-01527-y. PMID 34856928